CLINICAL TRIAL: NCT01012557
Title: H1N1v Vaccination of Pregnant Women: A Longitudinal Cohort Study Characterizing Influenza AH1N1v Vaccination in Pregnant Women
Brief Title: H1N1v Vaccination of Pregnant Women: A Longitudinal Cohort Study Characterizing Influenza A H1N1v Vaccination in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Studies on Asthma in Childhood (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H1N1v
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: H1N1v Influenza
Keywords: H1N1v; vaccine; pregnant; women; Assess whether the adjuvanted vaccine offers a meaningful benefit in pregnant women in terms of immune response over the non-adjuvanted vaccine.; Assess the persistence of immune response over a 15 month time period after one single vaccination of the pregnant mother.; Assess whether the immune response to H1N1 in pregnant women is different from that of non-pregnant women of similar age.; Gain insight on safety of the Novartis egg-based MF59 adjuvanted H1N1 vaccine Focetria in pregnant women and their babies.; Assess the maternally transferred specific antibodies against H1N1v in the newborn; Passive immunity transferred to the infant.
MeSH Terms: interventions — focetria

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pregnant women (>20 weeks), 7.5 mcg H1N1v full MF59 adjuvant (Active Comparator)
  Interventions: Biological: Focetria
- Pregnant women (>20 weeks), 3.75 mcg H1N1v half MF59 adjuvant (Active Comparator)
  Interventions: Biological: Focetria
- Pregnant women (>20 weeks), 15 mcg H1N1v unadjuvanted (Active Comparator)
  Interventions: Biological: Focetria
- Non-pregnant mothers, 7.5 mcg H1N1v full MF59 adjuvant (Active Comparator)
  Interventions: Biological: Focetria

INTERVENTIONS:
Biological: Focetria — 7.5 mcg H1N1v full MF59 adjuvant i.m.(intramuscular)x 1
  Arms: Pregnant women (>20 weeks), 7.5 mcg H1N1v full MF59 adjuvant
Biological: Focetria — 3.75 mcg H1N1v half MF59 adjuvant i.m.(intramuscular)x 1
  Arms: Pregnant women (>20 weeks), 3.75 mcg H1N1v half MF59 adjuvant
Biological: Focetria — 15 mcg N1N1v unadjuvanted i.m.(intramuscular) x 1.
  Arms: Pregnant women (>20 weeks), 15 mcg H1N1v unadjuvanted
Biological: Focetria — 7.5 mcg H1N1v full MF59 adjuvant i.m.(intramuscular) x 1
  Arms: Non-pregnant mothers, 7.5 mcg H1N1v full MF59 adjuvant

SUMMARY:
Pregnant women are at particular risk during the imminent H1N1v influenza pandemic. The new H1N1v virus requires urgent political and medical decisions on vaccination strategies in order to minimize severe disease and death from this pandemic. However, there is a lack of evidence to build such decisions upon. A vaccine will be provided in the fourth quarter of 2009, but there is little knowledge on the immunogenicity. Particularly its clinical effectiveness and duration of immunity in pregnant women and their newborn infants is unknown. Therefore, it will be important to study the optimal vaccination regimens with respect to dosing and use of adjuvant to decide future health policies on vaccination of pregnant women. We have a unique possibility to study these aspects of H1N1v infection in pregnant women in our ongoing unselected, prospective, birth-cohort study recruiting 800 pregnant mothers between Q1- 2009 and Q4-2010. Pregnant women from East-Denmark are being enrolled during the 2nd trimester and their infant will undergo a close clinical follow-up. The H1N1v pandemic is expected to reach Denmark Q4-2009. The timing of this enrollment and the imminent pandemic allows for an "experiment of nature" whereby the first half of the mothers completes pregnancy before the H1N1v pandemic. The other half of this cohort will be pregnant while H1N1v is prevalent in the community and will require H1N1v vaccination. The aim of this randomized, controlled, trial is to compare and evaluate the dose-related immune protection conferred by vaccine and adjuvant (Novartis vaccine Focetria) in pregnant women and non-pregnant women. In addition the protocol will assess the passive immunity conferred to the newborn from these vaccine regimes. The study will provide evidence-based guidance for health policies on vaccination for the population of pregnant women during future H1N1v pandemics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant and non pregnant women living in Eastern Denmark
* Fluent in Danish

Exclusion Criteria:

* Heart disease, endocrine disease, tuberculosis and sarcoidosis.
* History of any anaphylaxis, serious vaccine reactions, or hypersensitivity to influenza viral proteins, to any excipients, and to eggs (including ovalbumin), and chicken proteins.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Day 22/Day 1, and at all the other relevant time points to assess persistence/Day 1 geometric mean ratio (GMR) of HI | Day 1, Day 22
Geometric mean HI titer (GMT) on Day 1, Day 22, and at all the other relevant time points to assess persistence. | Day 1, Day 22
Percentage of subjects achieving a seroconversion or a significant increase (defined as: HI ≥1:40 for subjects negative at baseline [<1:10]; a minimum 4-fold increase in HI titer for subjects positive at baseline [HI≥1:10]) | Day 1, Day 22
Percentage of subjects with a HI titer ≥1:40 (i.e. seroprotection) on Day 1, Day 22, and at all the other relevant time points to assess persistence | Day 1, Day 22

SECONDARY OUTCOMES:
The safety of the study vaccines will be assessed based on number of subjects exposed to study vaccines with reported selected adverse events per vaccine group. | 12 months
The outcomes of pregnancies will be categorized as normal, abnormal or therapeutic/elective termination | duration of pregnancy

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - COPSAC, Gentofte Municipality
  - Næstved Hospital, Pediatric Department, Næstved

REFERENCES:
- [Background] Bischoff AL, Folsgaard NV, Vissing NH, Birch S, Brix S, Bisgaard H. Airway mucosal immune-suppression in neonates of mothers receiving A(H1N1)pnd09 vaccination during pregnancy. Pediatr Infect Dis J. 2015 Jan;34(1):84-90. doi: 10.1097/INF.0000000000000529. PMID 25229268
- [Result] Bischoff AL, Folsgaard NV, Carson CG, Stokholm J, Pedersen L, Holmberg M, Bisgaard A, Birch S, Tsai TF, Bisgaard H. Altered response to A(H1N1)pnd09 vaccination in pregnant women: a single blinded randomized controlled trial. PLoS One. 2013 Apr 18;8(4):e56700. doi: 10.1371/journal.pone.0056700. Print 2013. PMID 23637733